CLINICAL TRIAL: NCT02899052
Title: A Phase 2, Open-Label, Multi-Center Study of Venetoclax in Combination With Carfilzomib and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Venetoclax in Combination With Carfilzomib and Dexamethasone in Participants With Relapsed or Refractory Multiple Myeloma (MM)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc; Onyx Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-538; 2019-004340-30 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Refractory myeloma; Relapsed myeloma; Relapsed or Refractory
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — carfilzomib; venetoclax; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Carfilzomib + Dexamethasone (Experimental): Part 1: Evaluate the safety and pharmacokinetic profiles while providing information to determine the appropriate doses of venetoclax and carfilzomib (VenKd) to be used in the VenKd combination in approximately 18 participants. The dose levels are Venetoclax 400 mg or 800 mg; Carfilzomib 20/27 mg/m2, 20/70 mg/m2, and/or 20/56 mg/m2; Dexamethasone 40 mg
  Part 2: Further evaluate the safety and efficacy profile of the VenKd combination selected after completion of Part 1 in approximately 22 additional participants. Participants may discontinue Kd but may continue receiving venetoclax once daily (QD) as monotherapy.
  Part 3: Further evaluation of the efficacy of the VenKd combination after completion of Part 1 and Part 2 in 7 additional participants.
  Part 4, An additional 65 participants t(11;14) positive will receive varying doses of the VenKd combination or carfilzomib and dexamethasone
  Interventions: Drug: Carfilzomib; Drug: Venetoclax; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib lyophilized administered intravenously as a 10 to 30 minute infusion in Cycles 1 and beyond within 30 minutes to 4 hours after dexamethasone dosing.
  Dose level 1 (K1) Cycle 1: 20 mg/m2 on Days 1 and 2, 27 mg/m2 on Days 8, 9, 15, and 16; Cycles 2 - 12: 27 mg/m2 on Days 1, 2, 8, 9, 15, and 16; Cycles 13 - 18: 27 mg/m2 on Days 1, 2, 15, and 16; Cycles 19 and beyond, for participants that have not previously transitioned to monotherapy: 27 mg/m2 on Days 1, 2, 15, and 16.
  Dose Level K2: Cycle 1: 20 mg/m2 on Day 1; 70 mg/m2 on Days 8 and 15 Cycles 2 - onward: 70 mg/m2 on Days 1, 8, and 15. Dose Level K3: Cycle 1: 20 mg/m2 on Days 1 and 2; 56 mg/m2 on Days 8, 9, 15, and 16.
  Cycles 2 - onward: 56 mg/m2 on Days 1, 2, 8, 9, 15, and 16.
  Other Names: Kyprolis
Drug: Venetoclax — Venetoclax tablet administered orally once daily during Cycles 1 - onward. Venetoclax dose level 1 (Ven1) 400 mg once daily, Ven2 800 mg once daily.
  Other Names: Venclexta; ABT-199
Drug: Dexamethasone — Dexamethasone tablet administered orally during Cycles 1 - onward. Dexamethasone dose level 1 (Dex1) 40 mg once weekly, Dex2 40 mg once weekly, Dex3 20 mg twice weekly.

SUMMARY:
A Phase 2, open-label, dose escalation study to evaluate the safety and efficacy of venetoclax in combination with carfilzomib-dexamethasone (Kd) in participants with relapsed or refractory MM and have received 1 to 3 prior lines of therapy.

Part 4 of this study is currently enrolling.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Collaborative Oncology Group (ECOG) performance score of less than or equal to 2.
* Documented relapsed or progressive Multiple Myeloma (MM) on or after any regimen or is refractory to the most recent line of therapy.
* Positive for translocation t(11;14) as determined by an analytically validated Fluorescent In Situ Hybridization (FISH) assay per central laboratory testing.
* Received prior treatment with at least 1 prior line of therapy for MM.
* Measurable disease on Screening per International Myeloma Working Group (IMWG) criteria.
* Meets absolute neutrophil count, platelet count, hemoglobin, liver and kidney function laboratory values within 2 weeks prior to first dose of study drug.

Exclusion Criteria:

* Has a pre-existing condition that is contraindicated including.

  * Non-secretory or oligo-secretory MM
  * Active plasma cell leukemia.
  * Waldenström's macroglobulinemia.
  * Primary amyloidosis.
  * POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
  * Active hepatitis B or C infection based on screening blood testing.
  * Known active Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
  * Significant cardiovascular disease.
  * Major surgery within 4 weeks prior to first dose.
  * Acute infections requiring antibiotic, antifungal or antiviral therapy within14 days prior to first dose.
  * Peripheral neuropathy ≥ Grade 3 or ≥ Grade 2 with pain within 2 weeks prior to first dose.
  * Uncontrolled diabetes or uncontrolled hypertension within 14 days prior to first dose.
  * Any other medical condition that, in the opinion of the Investigator, would adversely affect the participant's participation in the study.
* History of other active malignancies, including myelodysplastic syndrome (MDS), within the past 3 years prior to study entry Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | First dose of study drug through at least 30 days after end of treatment (approximately 2 years)
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Very Good Partial Response (VGPR) or Better Response Rate of VenKd in Participants with Relapsed or Refractory Multiple Myeloma (RRMM) as well as Those with t(11;14)-positive RRMM | First dose of study drug through at least 30 days after end of treatment (approximately 2 years)
  VGPR or better response rate is defined as the percentage of participants with documented VGPR or better based on IMWG criteria.
Objective Response Rate (ORR) of VenKd in Participants with Relapsed or Refractory Multiple Myeloma (RRMM) as well as Those with t(11;14)-positive RRMM | First dose of study drug through at least 30 days after end of treatment (approximately 2 years)
  ORR is defined as the percentage of participants with a documented PR or better based on IMWG criteria.
Complete Response (CR) or Better Rate of VenKd in Participants with Relapsed or Refractory Multiple Myeloma (RRMM) as well as Those with t(11;14)-positive RRMM | First dose of study drug through at least 30 days after end of treatment (approximately 2 years)
  Complete response or better rate is defined as the percentage of participants with documented CR or better based on IMWG criteria.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Response Rate in Participants with Relapsed or Refractory Multiple Myeloma and in a Subset of Participants with High B-cell lymphocyte-2 (BCL-2) Expression | Up to approximately 17 months
  VGPR or better response rate is defined as the proportion of participants with documented VGPR or better based on IMWG criteria.
Progression-free survival (PFS) in Participants with Relapsed or Refractory Multiple Myeloma and in a Subset of Participants with High B-cell lymphocyte-2 (BCL-2) Expression | Up to approximately 17 months
  PFS is defined as the number of days from the date of the first dose of study drug to the date of the first documented progressive disease (PD) or death due to any cause, whichever occurs first.
Minimal residual disease (MRD) | Up to 2 years (Screening, Cycle 3 Day 1, and Confirmation of Stringent Complete Response [sCR]/Complete Response [CR])
  MRD in the bone marrow by next generation sequencing.
Duration of Overall Response (DOR) in Participants with Relapsed or Refractory Multiple Myeloma and in a Subset of Participants with High B-cell lymphocyte-2 (BCL-2) Expression | Up to approximately 17 months
  DOR is defined as the number of days from the participant's date of first documented response (PR or better) to the date of first documented PD or death due to MM, whichever occurs first.
Time to progression (TTP) in Participants with Relapsed or Refractory Multiple Myeloma and in a Subset of Participants with High B-cell lymphocyte-2 (BCL-2) Expression | Up to approximately 17 months
  TTP is defined as the number of days from the date of the first dose of study drug to the date of first documented PD or death due to MM, whichever occurs first.
Objective response rate (ORR) in Participants with Relapsed or Refractory Multiple Myeloma and in a Subset of Participants with High B-cell lymphocyte-2 (BCL-2) Expression | Up to approximately 17 months
  ORR is defined as the proportion of participants with documented partial response (PR) or better based on International Myeloma Working Group (IMWG) criteria.
Time to Response (TTR) in Participants with Relapsed or Refractory Multiple Myeloma and in a Subset of Participants with High B-cell lymphocyte-2 (BCL-2) Expression | Up to approximately 17 months
  TTR is defined as the number of days from the date of the first dose of study drug to the date of first documented response (Partial Response (PR) or better).
Area under the plasma concentration-time curve from 0 to 24 hours (AUC0-24) post-dose of Venetoclax | Approximately 24 hours post-dose on Cycle 1 Days 1 and 15
  AUC0-24 post-dose of venetoclax.
Clearance (CL) of Carfilzomib | Approximately 4 hours post-dose on Cycle 1 Days 1 and 15
  CL of carfilzomib.
Terminal Phase Elimination Rate Constant (β) of Carfilzomib | Approximately 4 hours post-dose on Cycle 1 Days 1 and 15
  β of carfilzomib.
AUC from 0 to Infinity (AUC∞) of Carfilzomib | Approximately 4 hours post-dose on Cycle 1 Days 1 and 15
  AUC∞ of carfilzomib.
AUC from Time 0 to the Time of the Last Measurable Concentration (AUCt) of Carfilzomib | Approximately 4 hours post-dose on Cycle 1 Days 1 and 15
  AUCt of carfilzomib.
Maximum Plasma Concentration (Cmax) of Venetoclax | Approximately 24 hours post-dose on Cycle 1 Days 1 and 15
  Cmax of venetoclax.
Cmax of Carfilzomib | Approximately 4 hours post-dose on Cycle 1 Days 1 and 15
  Cmax of carfilzomib.
Terminal Elimination Half-life (t1/2) of Carfilzomib | Approximately 4 hours post-dose on Cycle 1 Days 1 and 15
  t1/2 of carfilzomib.
Time to Maximum Plasma Concentration (Peak Time, Tmax) of Venetoclax | Approximately 24 hours post-dose on Cycle 1 Days 1 and 15
  (Peak time, Tmax) of venetoclax.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (32):
- United States (18):
  - University of Alabama at Birmingham - Main /ID# 151405, Birmingham, Alabama
  - University of Arkansas for Medical Sciences /ID# 151399, Little Rock, Arkansas
  - Memorial Healthcare System /ID# 224862, Hollywood, Florida
  - Winship Cancer Institute of Emory University /ID# 161710, Atlanta, Georgia
  - The University of Chicago Medical Center /ID# 151395, Chicago, Illinois
  - Indiana Blood & Marrow Transpl /ID# 218862, Indianapolis, Indiana
  - Duplicate_University of Kentucky Chandler Medical Center /ID# 151407, Lexington, Kentucky
  - Central Maine Medical Center /ID# 218856, Lewiston, Maine
  - Duplicate_University of Maryland School of Medicine /ID# 159721, Baltimore, Maryland
  - Oncology Hematology Associates (OHA) - Springfield /ID# 218855, Springfield, Missouri
  - Washington University-School of Medicine /ID# 222651, St Louis, Missouri
  - Duke Cancer Center /ID# 162062, Durham, North Carolina
  - University of Pennsylvania /ID# 151768, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center /ID# 218336, Dallas, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 218252, Temple, Texas
  - University of Utah /ID# 151397, Salt Lake City, Utah
  - Duplicate_VA Puget Sound Healthcare Syst /ID# 155369, Seattle, Washington
  - Aurora Health Care, Aurora Cancer Center /ID# 209612, Wauwatosa, Wisconsin
- Australia (4):
  - Border Medical Oncology Research Unit Albury Wodonga Regiona /ID# 222200, East Albury, New South Wales
  - Calvary Mater Newcastle /ID# 218739, Waratah, New South Wales
  - Flinders Medical Centre /ID# 221345, Bedford Park, South Australia
  - Royal Hobart Hospital /ID# 217546, Hobart, Tasmania
- Hungary (4):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 217624, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem /ID# 217626, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 217625, Budapest
  - Szegedi Tudományegyetem /ID# 219172, Szeged
- Puerto Rico (2):
  - Auxilio Mutuo Cancer Center /ID# 157853, San Juan
  - VA Caribbean Healthcare System /ID# 157854, San Juan
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol /ID# 218006, Badalona, Barcelona
  - Hospital Clinic de Barcelona /ID# 218007, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 218005, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 220925, Madrid

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Badawi MA, Engelhardt B, Dobkowska E, Deng R, Kaufman JL, Menon R, Salem AH. Exposure-response relationships of venetoclax in combination with carfilzomib and dexamethasone in relapsed/refractory t(11;14) multiple myeloma patients. Invest New Drugs. 2024 Dec;42(6):635-643. doi: 10.1007/s10637-024-01471-x. Epub 2024 Oct 10. PMID 39388024
- [Derived] Costa LJ, Davies FE, Monohan GP, Kovacsovics T, Burwick N, Jakubowiak A, Kaufman JL, Hong WJ, Dail M, Salem AH, Yang X, Masud AA, Munasinghe W, Ross JA, Bueno OF, Kumar SK, Stadtmauer EA. Phase 2 study of venetoclax plus carfilzomib and dexamethasone in patients with relapsed/refractory multiple myeloma. Blood Adv. 2021 Oct 12;5(19):3748-3759. doi: 10.1182/bloodadvances.2020004146. PMID 34470049